CLINICAL TRIAL: NCT06248957
Title: SYSTEMS-LEVEL ANALYSES OF IMMUNE DYSREGULATION
Acronym: SAID
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other); Uppsala University Hospital (Other); Region Halland (Other); Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Petter Brodin, M.D., Ph.D., Professor, Karolinska Institutet
Other Study IDs: 2023-06579-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Immunodeficiency; Autoimmune Diseases; Autoinflammatory Syndrome; Allergy; Dysregulated Host Response
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Autoimmune Diseases; Hypersensitivity | interventions — Immunomodulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with viable cells, DNA, plasma proteins. Microbiome samples from stool, airways and skin. Fibroblasts in selected cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with immune dysregulation: Patients sampled before and during different immunomodulatory therapies due to immune system dysregulation.
  Interventions: Combination Product: Immunomodulation
- Healthy subjects: Age-matched healthy individuals sampled longitudinally

INTERVENTIONS:
Combination Product: Immunomodulation — Variable protocols for combined immunomodulatory therapies currently in use for different forms of immune dysregulation
  Groups: Patients with immune dysregulation

SUMMARY:
The aim of the SAID study is to create a national resource in Sweden to enable comprehensive immunological analyses of an extremely complex and clinically challenging group of individuals with variable forms of immune system dysregulation. We hope to establish a biobank of primarily blood and fecal samples from children and adults, with confirmed or suspected immune dysregulation, as well as age- and sex- matched healthy controls, for comparisons of immune cell/mediator alongside various clinical presentations of these immunological diseases as well as microbiome samples as possible a possible modifier of clinical presentations. The project will also include the establishment of a national database with deep immunological data, treatment and clinical outcomes for these patients, accessible to participating researchers and clinicians.

DETAILED DESCRIPTION:
BACKGROUND

Immune dysregulation encompasses multiple different conditions in which the immune system does not function properly and displays inappropriate or inadequate responses, overreactions or under-reactions directed towards external or internal targets. It is a broad term, and its manifestations include several different categories of disease:

Immunodeficiencies: These disorders impair the immune system's ability to defend the body against foreign or abnormal cells that invade or attack it (such as bacteria, viruses, fungi, and cancer cells). As a result, unusual bacterial, viral, or fungal infections or lymphomas or other cancers may develop. Primary immunodeficiencies (PIDs) comprise a group of nearly 500 inherited disorders, often due to single-gene mutations that result in the specific impairments in immune function. Secondary immunodeficiencies (SIDs) involve a weakened immune system caused by external sources e.g. chemical (chemotherapy), infection (HIV) or cancer.

Autoimmune Disorders: In these conditions the production of autoantibodies against self-antigens causes the immune system to attack healthy cells and tissues. Some of the most common examples include type 1 diabetes (T1D), rheumatoid arthritis (RA), multiple sclerosis (MS), systemic lupus erythematosus (SLE).

Autoinflammatory Disorders: Here dysregulation of the innate immune system leads to spontaneous and recurrent inflammatory episodes. In contrast to autoimmune diseases where antibodies against self-antigens play a central role, the defect in autoinflammatory diseases often lies in the first responder, innate, arm of the immune system where the defect triggers inappropriate activation of the normal inflammatory response or disables resolution thereof. Examples include familial Mediterranean fever (FMF) and cryopyrin-associated periodic syndromes.

Severe allergies: Allergic reactions are misdirected reactions of the immune system to substances commonly found in the environment. Allergens elicit a T helper 2 immune response, including the involvement of IgE, mast cells, innate lymphoid cells 2 (ILC2), eosinophils, and basophils. Severe Allergy which does not respond to therapy can also indicate underlying immundysregulation.

Lymphoproliferation: Lymphoproliferation (LP) refers to persistent polyclonal, oligoclonal, or monoclonal proliferation of lymphoid cells in the clinical setting of immune dysregulation. Symptoms are non-specific and mimic those of an infection, inflammation, or neoplasia and are characterized by chronic or recurrent lymphadenopathy, hepatosplenomegaly, extranodal infiltration, and/or peripheral blood lymphocytosis. Immune disorders characterized by LP include autoimmune lymphoproliferative syndrome (ALPS) and X-linked lymphoproliferation (XLP).

Attempting to classify and group disorders of immune dysregulation in this way is of course an over-simplification as exemplified by conditions with both autoimmune and autoinflammatory components, such as psoriasis or IBD. For this reason, it has been proposed that manifestations of immune dysregulation should be considered as a continuum with rare monogenic autoimmune disorders at one end, rare monogenic autoinflammatory disorders at the other end, followed by polygenic autoimmune/autoinflammatory conditions respectively, with mixed pattern diseases in the center. In real life, patients with immune dysregulation also often present with more than one disease manifestation which further complicates diagnosis and treatment.

Finally, another factor that must be considered when trying to understand immune dysregulation, is the influence of the microbiome. Disruptions to the microbiota early in life are known to have lasting health effects, including increased risks of immune- mediated diseases such as allergy. However, less is known about the possibility that inborn errors of immunity may also shape the developing microbiome with ensuing health-related consequences, although the role of the microbiome in immune dysfunction is beginning to be appreciated. For example, impaired immunity may alter the intestinal microbiome causing subsequent increased intestinal permeability, with increased exposure to bacterial DNA and an activation of innate and adaptive immune that ultimately perpetuate or exacerbate any defects in immunity.

THE PROBLEM Certain types of immune dysregulation can be extremely rare and diagnosis and appropriate treatment are complicated issues. Some are caused by specific genetic mutations with on average one new genetic mutation associated with immune dysregulation being discovered every month. However, in over half of patients with e.g. autoinflammatory disorders, no genetic cause can be found. Some disorders also affect multiple branches of the immune system due to a broader inappropriate immune response, where signs and symptoms of autoimmunity, allergy, and/or immunodeficiency can all be present in one condition at the same time. A new approach is therefore essential to facilitate diagnosis and personalized treatment of patients with immune dysregulation which we believe will involve more holistic, systems-level analyses of immune cell composition and functional responses. Furthermore, little is known about the interaction between the immune function and microbiome composition, particularly in relation to immune dysregulation, and understanding this interplay may reveal new therapeutic opportunities and enable prediction of adverse outcomes.

SYSTEMS IMMUNOLOGY The human immune system consists of many specialized cell populations that stimulate each other to respond, but also compete for growth factors and directly suppress each other to prevent immune pathology. In this way the whole system functions as a highly integrated network. Since this network is decentralized without any master regulator, all actions in the system, both productive immune responses to microbes and destructive autoimmune attacks on normal tissues, emerge from the combined actions of the many immune cell populations that make up this network. To understand higher order functions in a system this complex, comprehensive analyses involving all cell populations simultaneously are required. Only then can the consequence of activating one, or a few specific cell populations, in the system as a whole be understood. This realization has led to the pursuit of "Systems Immunology", the application of technologies and theories from the field of Systems Biology to understand immune systems. Technological advances, primarily in mass cytometry for high- dimensional immune cell analysis, and high-throughput serum protein analyses, now allow for such detailed profiling of all components that make up human immune systems. We therefore now have the ability to dissect immune responses into their underlying cell-cell and cell-protein interactions.

SCIENTIFIC HYPOTHESIS

* Systems-level analyses of immune cell composition and functional responses can reveal distinct cellular networks and pathways related to immune dysregulation in patients with systemic inflammation and immune dysregulation of unknown cause, providing new targets for treatment and facilitating diagnosis.
* Inter-individual variation in systemic inflammatory diseases could be explained by differences in microbial colonization. We hypothesize that microbiome compositional differences can explain differences among patients with defects in similar immune system pathways.
* By combining systems-level functional analyses with whole genome sequencing (clinical analyses) we can better understand redundant pathways in human immune systems which modulate phenotypes in patients with systemic inflammatory and immune dysregulation diseases.

ELIGIBILITY:
Inclusion Criteria:

Patients of all ages seeking care or being referred for suspected immune dysregulation or with a known immune-mediated disease and failing to respond to standard therapy

Exclusion Criteria:

Healthy control individuals will be excluded on the basis of having a diagnosis of an immune mediated disorder, immunomodulatory treatment or current infection or cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects, children and adults in Sweden and referred to Swedish centers with known or suspected immune dysregulation.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
control of immune dysregulation | 1-3 months from start of therapy
  Remission and control of immune dysregulation manifested as reduced inflammation, symptom relieve and halted immunoproliferation for examples

SECONDARY OUTCOMES:
Exploratory immunological parameters | 1-3 months from start of therapy
  Systems-level immunomonitoring for exploration of cell state changes in response to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brodin lab website — https://www.brodinlab.com/